CLINICAL TRIAL: NCT05737901
Title: Effect of Different Discharge Training Methods On Readiness and Self-Efficacy for Discharge After Coronary Artery Bypass Surgery: A Randomized Uncontrolled Clinical Study
Brief Title: The Effect of Different Training Methods On Discharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Collaborators: Aydin Adnan Menderes University Member Training Program (Unknown); Aydın Adnan Menderes University Scientific Research Projects Unit (Unknown)
Responsible Party: Principal Investigator, Dilara ŞAHAN, Research assistant, PhD, Aydin Adnan Menderes University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AdnanU
Record Dates: First submitted 2023-01-31; First posted 2023-02-21 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Coronary Artery Bypass Graft; Discharge Education
Keywords: mobile applications; education; self efficacy; discharge readiness; coronary artery bypass; nursing

STUDY DESIGN:
Intervention Model Description: The study was carried out quasi-experimentally.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard care group (No Intervention): The standard discharge training of the clinic was carried out in the patient's room on the day of discharge in an average of 5 minutes, in the form of verbally explaining the information deemed important by the physician and/or nurse to the patient. No intervention was made in this group.
- Education Booklet Group (Experimental): Discharge training was given by the researcher the day before the surgery in an average of 60 minutes in the meeting room of the clinic through the booklet.
  Interventions: Other: Education Booklet
- Mobile Application Group (Experimental): The mobile application was introduced to the patient by the researcher the day before the surgery. During the presentation phase, the patient was informed about the titles and contents of the training videos, and after explaining the technical features related to turning the tablet on and off, raising and lowering the volume, logging into the account using the username and password for training, using the buttons on the main screen and the keyboard, the patient was asked to apply them. All these stages took an average of 20 minutes. In addition, information about logging in, such as how to switch on and off the device, the patient's user name and password, were added to the back of the tablet in writing.
  Interventions: Other: Mobile application

INTERVENTIONS:
Other: Education Booklet — Training titles and contents were created by listing the most common complications and needs of patients after CABG surgery. In the "General Information" section of the booklet, the definition of CAD, how CABG surgery is performed, the length of hospital stay, and what can be experienced in the hospital after surgery and in the home environment after discharge were discussed. In the "Postoperative Self-Care Practices" section, information about the healing process of the breastbone, pain management, medication, respiratory exercises, early nutrition, personal hygiene, protection from coronavirus-19, pulse control, postoperative heart attack, conditions to be reported, compression stockings use for varicose veins, physical activity, travel, sleep and rest, sexual life, and coping with stress and depression was presented. In the "Postoperative Life" section, training topics on exercise, nutrition, smoking, and alcohol use were included.
  Arms: Education Booklet Group
Other: Mobile application — The logo and content of the "Bypass e-Discharge" application was visually designed, and the software was developed. In-app transactions were secured with end-to-end encryption by entering the username and password, and internet access was not required to use the application. The application was presented for expert opinion (3 patients, 1 academician, 2 nurses, 2 physicians) in order to investigate the user experience, and edits were made on its interface (such as adding the "acceleration" feature in videos, an additional button for stopping and starting videos, displaying video total time on the screen, and magnification of all buttons).
  Arms: Mobile Application Group

SUMMARY:
This study was conducted to examine the effects of different discharge training methods on readiness to discharge and self-efficacy in individuals undergoing coronary artery bypass graft surgery.

DETAILED DESCRIPTION:
With the shortening of the length of hospital stay after coronary artery bypass graft (CABG) surgery, patients can be discharged by taking on complex responsibilities before the healing process is completed and before their perception of self-efficacy increases. Today, in the discharge training traditionally given with oral or written materials after surgery, the subjects that are generally considered important are selected, which may lead to not addressing the specific needs of individuals. In addition, inconsistencies may occur due to the trainer, too much written information that is beyond the knowledge level of the patients, frequent forgetting or incorrect remembering of the information given, and the incompatibility between the time planned by the nurse for the training and the time the patient feels ready. In one study, it was reported that 55.3% of the nurses did not provide patient education, education was in the seventh place in their daily work routines, and the reasons for not training the patients were their excessive workload and inability to use time effectively. For this reason, traditional patient education methods have begun to be replaced by technological methods. Mobile applications create opportunities for patients to participate in their own care during their hospital stay in the remaining time spent on examinations and treatments. It has been reported that video interventions are extremely effective, especially in populations with low literacy rates, and longer-term information transfer can be achieved by leaving tablets used for educational purposes in the patient room.

CABG surgery is most needed during middle and advanced ages. However, it is generally known that elderly individuals are mostly not familiar with recent mobile technologies. In Turkey, no research has been found on whether this patient group is suitable for using mobile technologies, the effectiveness of tablets in providing information to inpatients, the extent to which patients are interested and engaged with the application, the effectiveness of the application to bring the patient to a readiness state for discharge, the effect of the application on the perception of self-efficacy, and how it affects the state of satisfaction. Some authors also state that well-designed and reported studies are needed to demonstrate the effectiveness of mobile phone or tablet-based applications in the management of CAD (Coronary Artery Disease).

ELIGIBILITY:
Inclusion Criteria:

* Being literate
* Understanding and speaking the Turkish language
* Having undergone a planned open-heart surgery for the first time.

Exclusion Criteria:

* Patients who received psychiatric diagnosis
* Who were unable to use the tablet and mobile application after explanations
* Who had postoperative hospitalization for more than 10 days
* Who had a development of disorientation in the postoperative service
* Who had a valve surgery added to their CABG surgery during the operation were excluded from the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Barnason Efficacy Expectation Scale (BEES) - Cardiac Surgery Version | on the day of discharge after standard care, estimated average 7 days and one month after discharge
  The increasing score indicates that the individual's expectation of self-efficacy regarding recovery and behavioral changes is also high.
Readiness for Hospital Discharge Scale | on the day of discharge after standard care, estimated average 7 days
  The patient with a ready-to-discharge score of 7 and above is considered ready to be discharged, whereas a score below 7 indicates that the patient is not ready.

SECONDARY OUTCOMES:
System Usability Scale (SUS) | on the day of discharge after standard care, estimated average 7 days
  The increasing score indicates that the usability of the developed system has increased
Net Promoter Score | on the day of discharge after standard care, estimated average 7 days
  People who respond with a score of 9 or 10 are labeled as 'promoters,' those who receive a score of 7 or 8 are labeled as 'neutrals,' and those who score 6 or less are labeled as 'detractors.'

CONTACTS AND LOCATIONS:
Overall Officials: Dilara ŞAHAN, PhD, Principal Investigator — Aydin Adnan Menderes University
Locations (1):
- Aydın Adnan Menderes University, Aydin, Merkez, Turkey (Türkiye)

REFERENCES:
- [Result] Cook DJ, Moradkhani A, Douglas KS, Prinsen SK, Fischer EN, Schroeder DR. Patient education self-management during surgical recovery: combining mobile (iPad) and a content management system. Telemed J E Health. 2014 Apr;20(4):312-7. doi: 10.1089/tmj.2013.0219. Epub 2014 Jan 20. PMID 24443928
- [Result] Greysen SR, Khanna RR, Jacolbia R, Lee HM, Auerbach AD. Tablet computers for hospitalized patients: a pilot study to improve inpatient engagement. J Hosp Med. 2014 Jun;9(6):396-9. doi: 10.1002/jhm.2169. Epub 2014 Feb 13. PMID 24523051
- [Result] Noor Hanita Z, Khatijah LA, Kamaruzzaman S, Karuthan C, Raja Mokhtar RA. A pilot study on development and feasibility of the 'MyEducation: CABG application' for patients undergoing coronary artery bypass graft (CABG) surgery. BMC Nurs. 2022 Feb 4;21(1):40. doi: 10.1186/s12912-022-00814-4. PMID 35120517
- [Result] van Steenbergen GJ, van Veghel D, Ter Woorst J, van Lieshout D, Dekker L. IMPROV-ED trial: eHealth programme for faster recovery and reduced healthcare utilisation after CABG. Neth Heart J. 2021 Feb;29(2):80-87. doi: 10.1007/s12471-020-01508-9. Epub 2020 Nov 3. PMID 33141398